CLINICAL TRIAL: NCT07375888
Title: The Application of an Innovative Reactive Agility Testing System for Assessment in Older Adults With Dynapenia
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Fan-Chen Liu, Principal Investigator, Kaohsiung Medical University
Other Study IDs: KMUHIRB-E(I)-20250028; KMUHIRB-E(I)-20250028 (Other: Kaohsiung Medical University Chung-Ho Hospital Institutional Review Board)
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dynapenia
Keywords: Dynapenia; Elderly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Elderly: Normal muscle mass Normal muscle strength Normal physical performance
  Interventions: Diagnostic Test: Reactive Agility Testing System
- Pre sarcopenia: Low muscle mass Normal muscle strength Normal physical performance
  Interventions: Diagnostic Test: Reactive Agility Testing System
- Sarcopenia: Low muscle mass Low muscle strength or low physical performance
  Interventions: Diagnostic Test: Reactive Agility Testing System
- Dynapenia: Normal muscle mass Low muscle strength or low physical performance
  Interventions: Diagnostic Test: Reactive Agility Testing System

INTERVENTIONS:
Diagnostic Test: Reactive Agility Testing System — The participant stands in the preparation area located at the center of the testing field, which measures 1 m × 1 m. One sensor light is placed on each side, with each light positioned 3 meters away from the preparation area.
  After the system is activated, one of the lights will illuminate randomly between 1 and 5 seconds. Once the light turns on, the participant moves forward quickly, passes through a photo gate next to the preparation area, and continues forward until touching the sensor light to turn it off.
  The system records the time from when the light turns on to when the participant passes through the photo gate, which is defined as the decision time. The time from passing through the photo gate to touching and turning off the sensor light is defined as the movement time.
  After completing five trials on each side, the test ends. Finally, the system calculates the total time, which is the sum of the decision time and movement time.

SUMMARY:
Before the experiment, the researchers explain the purpose and procedures to the participants. After signing the informed consent form and completing basic personal information, participants perform a 5-minute warm-up. They then practice the test procedure 1-3 times to become familiar with the visual stimuli, followed by a 3-minute rest before the formal experiment.

Body composition and physical performance are assessed using handgrip strength, the five-time sit-to-stand test, and the skeletal muscle mass index.

Fall risk is evaluated using a localized fall risk awareness questionnaire.

Agility is tested using a reaction-based running task. Participants stand in a 1 m × 1 m preparation area, and one of two sensor lights placed 3 meters away lights up randomly. Participants run forward, pass through a photo gate, and touch the light to turn it off. Decision time, movement time, and total time are recorded over 10 trials.

DETAILED DESCRIPTION:
Before the experiment begins, the researchers will first explain the experimental procedures and purpose to the participants. Participants will then complete an informed consent form and provide their basic personal information. After that, participants will perform a 5-minute warm-up exercise.

To familiarize participants with the visual stimuli, they will practice the test procedure one to three times. After the practice session, participants will rest for 3 minutes before the formal experiment begins.

* (1) Body Composition and Physical Performance Data

  * **Handgrip Strength:** Measured using a handgrip dynamometer. Three trials are performed, and the maximum value is recorded as the handgrip strength.
  * **Five-Time Sit-to-Stand Test:** The participant sits on a standard testing chair with the hips and knees flexed at 90 degrees. Without using the hands for assistance, the participant performs five sit-to-stand movements as quickly as possible. The completion time is recorded.
  * **Skeletal Muscle Mass Index (SMI):** The participant stands barefoot on the measurement device and holds the hand electrodes to obtain appendicular muscle mass. The appendicular muscle mass is then divided by height squared to calculate the skeletal muscle mass index.
* (2) Fall Risk

Fall risk is assessed using a localized Fall Risk Awareness Scale. A higher score indicates a greater risk of falling and a higher level of fear of falling.

### (3) Agility Test

The participant stands in the preparation area located at the center of the testing field, which measures 1 m × 1 m. One sensor light is placed on each side, each positioned 3 meters away from the preparation area.

After the system is activated, one of the lights will illuminate randomly between 1 and 5 seconds. Once the light turns on, the participant moves forward quickly, passes through a photo gate next to the preparation area, and continues forward until touching the sensor light to turn it off.

The system records:

* **Decision time:** the time from when the light turns on to when the participant passes through the photo gate.
* **Movement time:** the time from passing through the photo gate to touching and turning off the sensor light.

After a total of 10 trials (combined left and right sides), the test ends. Finally, the system calculates the **total time**, which is the sum of the decision time and movement time.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 65 years and above
* Able to communicate with the researchers through spoken or written language
* Able to cooperate with all required assessments

Exclusion Criteria:

* Individuals with cognitive impairment
* Individuals who experience chest pain during recent exercise
* Individuals with angina or joint pain
* Individuals with congestive heart failure
* Individuals who have been advised by a physician not to exercise
* Patients with cancer currently receiving chemotherapy or radiotherapy
* Individuals with neuromuscular disorders or musculoskeletal injuries involving the ankle, knee, or hip joints

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older adults aged 65 years and above Able to communicate with the researchers through spoken or written language Able to cooperate with all required assessments
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2025-11-24 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2025-12-24 (Actual)

PRIMARY OUTCOMES:
Decision time | From participant enrollment to the end of testing
  The system records the time from when the light turns on to when the participant passes through the photo gate, which is defined
movement time | From participant enrollment to the end of testing
  The time from passing through the photo gate to touching and turning off the sensor light

SECONDARY OUTCOMES:
Handgrip Strength | From participant enrollment to the end of testing
  Measured using a handgrip dynamometer. Three trials are performed, and the highest value is recorded as handgrip strength.
Five-Time Sit-to-Stand Test | From participant enrollment to the end of testing
  The participant sits on a standard testing chair with the hips and knees flexed at 90 degrees. Without using the hands for assistance, the participant performs five sit-to-stand movements as quickly as possible. The completion time is recorded.
Skeletal Muscle Mass Index (SMI) | From participant enrollment to the end of testing
  The participant stands barefoot on the measurement device and holds the hand electrodes to obtain appendicular muscle mass. The appendicular muscle mass is then divided by height squared to calculate the skeletal muscle mass index.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting information will be available starting 2 years after the publication of the primary study results and will remain accessible for 5 years.
Access Criteria: The related supporting documents will only be made available to qualified researchers affiliated with academic institutions, medical organizations, or public health agencies, Applicants must submit a detailed research proposal and ethical approval documents, and access will be granted only upon approval.